CLINICAL TRIAL: NCT07018596
Title: Safety and Effectiveness of the CellFX® nsPFA Catheter Endocardial Ablation System for the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: NS-PFA Catheter Ablation of Paroxysmal Atrial Fibrillation With the Pulse Biosciences CellFX System
Acronym: NANOPULSE-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-CCP-US-043
Record Dates: First submitted 2025-06-05; First posted 2025-06-12 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation Paroxysmal; Cardiac Ablation; Cardiac Arrhythmia
Keywords: nsPFA; Pulsed Field Ablation; nano-PFA
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- nsPFA Cardiac Catheter System Treatment Arm (Experimental): Nanosecond Pulsed Field Ablation (nsPFA) technology will be used for ablating cardiac tissue using the CellFX nsPFA Cardiac Catheter System
  Interventions: Device: CellFX nsPFA Cardiac Catheter System

INTERVENTIONS:
Device: CellFX nsPFA Cardiac Catheter System — The CellFX nsPFA Cardiac Catheter System includes the nsPFA 360 Endocardial Ablation Catheter, CellFX Console, switcher box/adapter, and sensing cable. The System is a proprietary endocardial catheter system designed for use in cardiac electrophysiology procedures to treat arrhythmias, including atrial fibrillation. The nano-PFA 360 Catheter ablates cardiac tissue using nonthermal nanosecond pulses of electrical energy. nsPFA is a cell-specific, nonthermal ablation technology that delivers nanosecond-duration pulses of high-amplitude electrical energy to tissue via bipolar electrodes. The pulses disrupt the cell's and internal organelles' ability to maintain cellular homeostasis by creating nanopores in lipid membranes, ultimately leading to regulated cell death (RCD).

SUMMARY:
The objective of this study is to demonstrate the safety and effectiveness of the CellFX nano-second Pulsed Field Ablation (nsPFA) Cardiac Catheter Ablation System in treating recurrent, drug-resistant, symptomatic paroxysmal atrial fibrillation (AF).

DETAILED DESCRIPTION:
This study is a prospective, multicenter, non-randomized clinical investigation. Eligible participants with drug-resistant paroxysmal AF who are clinically indicated for a cardiac catheter ablation procedure will undergo nsPFA ablation with the CellFX Cardiac Catheter Ablation System. The primary endpoints will be assessed at 6 months after the ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of recurrent drug-resistant symptomatic paroxysmal AF defined as AF that terminates spontaneously or with intervention within seven (7) days of onset, documented by the following:

  i. Physician's note indicating the presence of AF symptoms and at least two (2) episodes of self-terminating AF within six (6) months prior to enrollment
* Age 18 through 85 years old (or older than 18 if required by local law)
* Failure of at least one AAD (class I or III) for AF as evidenced by recurrence of symptomatic AF, or intolerable side effects due to AAD.
* Participant is willing and capable of providing Informed Consent
* Received a standard cardiac work up and is an appropriate candidate for an investigational procedure as determined by study investigators

Exclusion Criteria:

* Left atrial diameter ≥5.5 cm (anteroposterior)
* Any of the following within 3 months prior to enrollment:

  1. Any cardiac surgery
  2. Myocardial infarction
  3. Percutaneous Coronary Intervention (PCI) / Percutaneous Coronary Intervention (PTCA) or coronary artery stenting
  4. Unstable angina
  5. Pericarditis or symptomatic pericardial effusion
* Any of the following within 6 months prior to enrollment:

  1. Any cerebral ischemic event (stroke or transient ischemic attack (TIA)
  2. History of thromboembolic event
* Prior history of medical procedure involving instrumentation of the left atrium (previous ablation, atrial septal defect (ASD) closure, Left atrial appendage occlusion)
* Planned Left Atrial Appendage (LAA) closure procedure, Transcatheter Aortic Valve Replacement (TAVR), Mitraclip, Atrial Septal Defect (ASD) or Patent Foramen Ovale (PFO) closure, Triclip or implant of an Implantable Loop Recorder (ILR), permanent pacemaker, biventricular pacemaker, or any implantable cardiac defibrillator (with or without biventricular pacing function) during or for any time during the follow-up period
* Patient who is not on oral anticoagulation therapy for at least 3 weeks prior to the ablation procedure
* Documented left atrial (LA) thrombus by imaging within 48 hours of the procedure.
* Presence of a permanent pacemaker, biventricular pacemaker, or any type of implantable cardiac defibrillator (with or without biventricular pacing function).
* Prior diagnosis of pulmonary vein stenosis
* Valvular cardiac surgical/percutaneous procedure (e.g., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve).
* Moderate to severe mitral valve stenosis
* More than moderate mitral regurgitation (i.e., 3+ or 4+ MR)
* New York Heart Association (NYHA) Class III or IV congestive heart failure or documented left ventricular ejection fraction (LVEF) less than or equal to 35% measured by acceptable cardiac testing (e.g., TTE)
* History of pulmonary hypertension with pulmonary systolic artery pressure >50 mm Hg, severe Chronic Obstructive Pulmonary Disease or restrictive lung disease
* Rheumatic heart disease
* Contraindication to anticoagulation (i.e., Heparin, Dabigatran, Apixaban, Vitamin K Antagonists such as warfarin)
* Active systemic infection
* Hypertrophic or advanced infiltrative cardiomyopathy
* Atrial myxoma
* Known reversible causes of AF, including but not limited to uncontrolled hyperthyroidism, severe untreated obstructive sleep apnea, and acute alcohol toxicity
* History of abnormal bleeding and/or clotting disorder
* Renal insufficiency with an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
* History of severe chronic gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
* Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
* Any woman known to be pregnant or breastfeeding, or any woman of childbearing potential who is not on a reliable form of birth regulation method or abstinence
* Other criteria, which the Investigator determines would make the patient unsuitable to participate (e.g. uncontrolled drug and/or alcohol addiction, congenital disease, fragility)
* Body Mass Index (BMI) > 40.0
* Participants with any other significant uncontrolled or unstable medical condition (such as uncontrolled brady-arrhythmias, ventricular arrhythmias, hyperthyroidism or significant coagulation disorder)
* Life expectancy less than one year
* Current or anticipated participation in any other clinical study of a drug, device, or biologic during the duration of the study not pre-approved by the Sponsor
* Unwilling or unable to comply fully with study procedures and follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with freedom from primary safety endpoint | Within 7 days, 30 days, and 6 months post-ablation procedure
  The primary safety endpoint is freedom from a primary safety endpoint for the following:
  * Cerebrovascular accident/Stroke
  * Thromboembolism
  * Myocardial infarction
  * Severe Pericarditis (requiring intervention)
  * Transient ischemic attack
  * Vagal nerve injury resulting in esophageal dysmotility or gastroparesis
  * Major vascular access complications
  * Bleeding
  * Pulmonary edema
  * Heart Block
  * Permanent Phrenic Nerve paralysis
  * Device or Procedure-related Death
  * CellFX System-related or PFA procedure-related cardiovascular and/or pulmonary adverse event that prolongs or requires hospitalization for more than 48 hours, excluding recurrent atrial fibrillation/atrial flutter/atrial tachycardia (AF/AFL/AT)
  * Cardiac tamponade/perforation
  * Significant acute kidney injury secondary to hemolysis
  * Pulmonary vein stenosis
  * Esophageal perforating complications
Proportion of participants achieving freedom from treatment failure. | 6 months post-ablation
  Acute procedural failure is defined as the inability to isolate all targeted pulmonary veins (PV) (minimally assessed for entrance block and, where assessable, exit block) during the index procedure or PV ablation using a non-study device in the left atrium

SECONDARY OUTCOMES:
Proportion of participants achieving acute procedural success | Immediately post-ablation procedure
  Acute Procedural Success: Ability to isolate all pulmonary veins and no ablation using a non-study device in the left atrium.

CONTACTS AND LOCATIONS:
Overall Officials: David Kenigsberg, MD, Study Chair — Pulse Biosciences, Inc.
Locations (1):
- Na Homolce Hospital, Prague, Roentgenova, Czechia

IPD SHARING:
Plan to Share IPD: No